CLINICAL TRIAL: NCT04113993
Title: Bazedoxifene - A New Selective Estrogen Receptor Modulator Treatment for Women With Schizophrenia: a Double-blind, Randomized, Placebo Controlled Trial
Brief Title: Bazedoxifene -Treatment for Women With Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Alfred (Other)
Collaborators: Monash University (Other); Monash Health (Other)
Responsible Party: Principal Investigator, Jayashri Kulkarni, Professor, Director of Monash Alfred Psychiatry research centre, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HREC Reference 47262
Record Dates: First submitted 2019-06-26; First posted 2019-10-03 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Schizophreniform Disorders; Schizo Affective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — bazedoxifene

STUDY DESIGN:
Intervention Model Description: This randomized, double-blind, placebo-controlled, 12-week trial will be conducted at two sites- the lead site is the Monash Alfred Psychiatry research Centre in Melbourne (Investigator - Prof Jayashri KULKARNI) , and a second site in Melbourne - The Monash Medical Centre (Investigator - Prof Suresh Sundram). The trial will follow the parallel comparison design consisting of two arms over 12 weeks (treatment x time). Participants will be screened to ensure inclusion / exclusion criteria are met.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomised to receive either activie treatment or identically packaged placebo
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Bazedoxifene (Experimental): Oral Bazedoxifene dosed at 40 mg daily
  Interventions: Drug: Bazedoxifene Acetate
- Placebo (Placebo Comparator): Identically packaged placebo capsule daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bazedoxifene Acetate — Oral Bazedoxifene dosed at 40 mg daily for 12 weeks
  Arms: Oral Bazedoxifene
Drug: Placebo — Identically packaged placebo capsule daily
  Arms: Placebo

SUMMARY:
To study the effect of adjunctive bazedoxifene - a selective estrogen receptor modulator (SERM) in a double blind, placebo-controlled adjunctive study in the treatment of women with schizophrenia. All patients receive standardized antipsychotic medication.

DETAILED DESCRIPTION:
Despite advances in the treatment of schizophrenia, pharmacotherapy remains sub- optimal, and the prognosis for many patients is poor. We have pioneered work showing that estradiol has a positive role in the treatment of psychosis symptoms and cognitive deficits seen in people with schizophrenia. However, with the longer-term work from studies such as the Women's Health Initiative (1), it has become clear that long-term use of estradiol with progesterone may have associated increased risks of breast and other cancers. Hence, we began working with the Selective Estrogen Receptor Modulator - raloxifene, which appears to be safer for longer term use with respect to the development of breast and other cancers. Building on our and others work, raloxifene used as an adjunctive treatment in schizophrenia appears to produce inconsistent and varying responses in different sub-populations; gender, menopausal status, age, drug dose and delivery mode. We now propose to conduct a double-blind, randomized, placebo controlled trial of a third generation SERM - bazedoxifene - which is 4 times more selective for the alpha than the beta oestrogen receptor subtype. Bazedoxifene appears to be safer with respect to long term use than older SERMs, has additional actions on the glucocorticoid receptor, and together this different pharmacology speculatively has greater potential than other SERMs to impact favorably on both psychosis symptoms and cognition in men and women with schizophrenia. This study will test 160 women to determine if bazedoxifene, as an adjunctive hormone modulator, is effective for positive and cognitive symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Physically well.
* A current DSM-V diagnosis of schizophrenia or related disorder.
* 18- 65 years
* Able to give informed consent.
* PANSS total score between 40 and 90 and a score of 4 (moderate) or more on two or more of the following PANSS items: delusions, hallucinatory behaviour, conceptual disorganization or suspiciousness.
* Documented normal PAP smear and pelvic examination in the preceding two years.
* Stable psychotropic medication for previous 4 weeks
* Normal breast ultrasound
* IQ > 70 (as determined by the WAIS IV subtests)
* English language proficiency (in order to provide informed consent and complete cognitive test battery)

Exclusion Criteria:

* Patients with known abnormalities in the hypothalamo-pituitary gonadal axis, thyroid dysfunction, central nervous system tumours, active or past history of a venous thromboembolic event.
* Patients with a history of severe traumatic brain injury or significant neurological or unstable medical illness such as epilepsy and diabetes or known active cardiac, renal or liver disease; presence of illness causing immobilisation.
* Patients whose psychotic illness is directly related to illicit substance use or who have a history of substance dependence during the last six months (with the exclusion of caffeine and/or nicotine dependence).
* Women aged 40 or over who have not had a normal mammogram in the last 24 months
* Use of any form of estrogen, progestin or androgen as hormonal therapy in preceding 4 weeks including the pill.
* Pregnant (HCG will be measured at screening)
* Breastfeeding
* Planned changes to psychotropic medication or psychotherapy regimen.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 160 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Schizophrenia symptoms | 12 Weeks
  Symptoms of schizophrenia as measured on the Positive and Negative Symptom Scale (PANSS).
  Subscales: Positive, Negative, General Psychopathology.
  Positive scale: 7 Items, (minimum score = 7, maximum score = 49). Negative scale: 7 Items, (minimum score = 7, maximum score = 49). General Psychopathology scale:16 Items, (minimum score = 16, maximum score = 112).
  PANSS Total score (summed from subscales): minimum = 30, maximum = 210
  For all items, higher values indicate increased symptom severity.

SECONDARY OUTCOMES:
Cognition | 12 Weeks
  The neuropsychological battery will include subtests from the following batteries:
  MATRICS Consensus Cognitive Battery (MCCB) comprises 7 domains: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving and social cognition.
  The Repeatable Battery for Neuropsychological Status (RBANS) comprises 12 subtests that are used to calculate five index scores (Immediate Memory; Visuospatial/Constructional; Language; Attention and Delayed Memory) and a total score.
  A verbal fluency task (Controlled Oral Word Association Task; COWAT), visual attention task (Trails A and B) and measures of premorbid intellect (Test of Premorbid Functioning; TOPF) will also be included.
  Eye tracking will be an optional extra and will be recorded using The EyeLink (SR Research Ltd). Participants will fixate and/or shift their gaze in response to a number of stimuli, appearing on the screen, as requested by the assessor.

CONTACTS AND LOCATIONS:
Locations (1):
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia